CLINICAL TRIAL: NCT02312440
Title: Comparison of Topical and Intravenous Tranexamic Acid on Blood Loss and Transfusion Rates in Total Hip Arthroplasty
Brief Title: Comparison of Topical and Intravenous Tranexamic Acid in Total Hip Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, zhoukaidi, MD in Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JTU-GK-010
Record Dates: First submitted 2014-11-10; First posted 2014-12-09 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-05

CONDITIONS: Blood Loss
Keywords: tranexamic acid; blood loss; topical administration; intravenous administration
MeSH Terms: conditions — Hemorrhage | interventions — Sodium Chloride; Saline Solution; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group1 (Placebo Comparator): 60 Milliliters（ml）Normal saline (0.9% sodium chloride) will be applied by soaking the hip cavity for at least 3 minutes before wound closure and then sucked away.
  Interventions: Drug: 0.9% sodium chloride
- Group2 (Experimental): two-dose intravenous tranexamic acid will be applied as follow: 10mg/kg of Tranexamic Acid in 100 Milliliters（ml) normal saline (0.9% sodium chloride),the first dose 15' prior to skin incision and the second dose at 180' after the first dosage.
  Interventions: Drug: tranexamic acid
- Group 3 (Experimental): 3g Tranexamic Acid diluted to 60 Milliliters（ml） with normal saline (0.9% sodium chloride) will be applied by soaking the hip cavity for at least 3 minutes before wound closure and then sucked away.
  Interventions: Drug: tranexamic acid

INTERVENTIONS:
Drug: 0.9% sodium chloride — The normal saline solution will be prepared under sterile conditions. In the operation room the sterile bag containing the solution will be given to the scrub nurse. The contents (60 ml) will be emptied in a sterile surgical bowl and the nurse will ask the surgeon to apply the solution before wound closure.The dosage and applying route can also be looked up in doctor's order sheet.
  Other Names: normal saline
  Arms: Group1
Drug: tranexamic acid — The Tranexamic Acid solution will be prepared under sterile conditions. In the operation room the sterile bag containing the solution will be given to the scrub nurse. The contents (60 ml) will be emptied in a sterile surgical bowl and the nurse will ask the surgeon to apply the solution before wound closure.The dosage and applying route can also be looked up in doctor's order sheet.
  Other Names: Cyclokapron
  Arms: Group2
Drug: tranexamic acid — The Tranexamic Acid solution will be prepared under sterile conditions. In the operation room the sterile bag containing the solution will be given to the circuit nurse and the circuit nurse will ask the anesthetist to apply the solution intravenously before tourniquet deflation. The dosage and applying route can also be looked up in doctor's order sheet.
  60 Milliliters（ml） by irrigation for 3 minutes before wound closure.
  Other Names: Cyclokapron
  Arms: Group 3

SUMMARY:
Recently, there has been interest in applying tranexamic acid topically before the closure of surgical wounds in total hip replacement. It has the advantages of ease of application, maximum concentration at the site of bleeding, minimising its systematic absorption and, potentially , decline the risks for systematic side-effects 。

DETAILED DESCRIPTION:
Objectives:To assess the efficacy and safety between the two different applying routes.

Patients in this project are randomly divided into three groups , one group is a blank group and the rest two groups receive either the topical or the intravenous form of tranexamic acid during unilateral THA(total hip arthroplasty).The total blood loss(TBL) will be calculated as the primary outcome for efficacy while the events of Deep Vein Thrombosis、Pulmonary Embolism、Acute Myocardial Infarction 、 Acute Kidney Infarction and Cerebral Infarction will be recorded to assess the safety of the tranexamic acid during a six-week follow-up for each patient.

All surgery are under general anesthesia, through direct lateral approach with cementless prosthesis. For all patients, the drain tube is clamped and closed completely for 2 hours; then the clamp is fully opened.

ELIGIBILITY:
Inclusion Criteria:

1. Consented to join in our project.
2. Adult patients (greater than 18 years old)
3. Patients scheduled for primary unilateral hip arthroplasty Patients for Ruijin hospital, Shanghai, China

Exclusion Criteria:

1. Patients who refuse to sign the Inform Consent
2. Had an allergy to TXA.
3. long-term bed >=3 weeks.
4. Using anticoagulant drugs within a week.
5. Coagulopathy (preoperative platelet count <150,000/mm3, INR>1.4, prolonged Activated Partial Thromboplastin Time，Prothrombin Time ，or thrombin time (>1.4 times longer than normal)
6. Pregnancy
7. Breastfeeding
8. Major comorbidities: Severe ischemic heart disease(class III and IV of New York Heart Association); sleep apnea syndrome; renal dysfunction ( glomerular filtration rate<60); or hepatic disfunction(glutamic-pyruvic transaminase>80 or glutamic oxalacetic transaminase>80).Retinopathy (disturbances of color vision).
9. History of thromboembolic disease: .
10. Been participating or been participated within a year in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Total Blood Loss（TBL） | estimated by an equation at the fifth postoperative day
  Total Blood Loss（TBL） was estimated with equations described by Gross et al.

SECONDARY OUTCOMES:
Transfusion rates | from the day of surgery to the day of discharge,an expected average of 7 days
  Include The number of units of perioperative blood transfusions, both intraoperative and postoperative, over the course of the patient's hospital stay
Venous thromboembolic event (symptomatic deep vein thrombosis or pulmonary embolism) | twelve weeks after surgery
  Clinically proven symptomatic deep vein thrombosis (DVT) or pulmonary embolism (PE)
other thromboembolic event | twelve weeks after surgery
  Clinically proven Acute Myocardial Infarction 、 acute kidney infarction or cerebral infarction
drainage output | ti will be recorded at the first day and the second day after surgery
  The amount of blood collected by a drain attached to the hip is measured 48 hours after surgery

OTHER OUTCOMES:
length of incision leakage | at the every day until the leakage stop,an expected average of 5 days
  patients will not be allowed to leave the hospital until the leakage stoped
Disseminated Intravascular Coagulation（DIC） | at any day before surgery and the first the fifth day after surgery
  include Activated Partial Thromboplastin Time（APTT）；Thrombin Time(TT) Prothrombin Time（PT);International Normalized Ratio(INR);Fibrinogen(FG); Fibrin degradation products(FDPs) D-Dimer
ecchymosis area | at the seventh day after surgery
  the investigators use the percentage of body surface area to record this outcome
human serum albumin | from the day of surgery to the day of discharge,an expected average of 7 days
  the investigators record the dosage of the human blood albumin used in each group.
American Society of Anesthesiologists Physical Status Classification (ASA class) | at the day of surgery
  the investigators record ASA class of every patients in each group.

CONTACTS AND LOCATIONS:
Overall Officials: jianmin feng, master, Principal Investigator — ruijin hospital，shanghai
Locations (1):
- Orthopedic Department of Ruijin hospital, Shanghai, Shanghai Municipality, China